CLINICAL TRIAL: NCT04556812
Title: Adults Habitual Patellar Dislocation:a Multiple-center Clinical Investigation Regarding Diagnosis and Therapeutic Strategy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hui Zhang (Other)
Responsible Party: Sponsor-Investigator, Hui Zhang, Doctor of Sports Medicine Service of Beijing Jishuitan hospital, Beijing Jishuitan Hospital
Organization: Beijing Jishuitan Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HuiZ-2
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Habitual Patellar Dislocation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): underwent "four-in-one" surgical technique centered on "tibial tuberosity osteotomy and proximal displacement"
  Interventions: Procedure: Four-in-one procedure
- Control group (Placebo Comparator): traditional soft tissue surgery
  Interventions: Procedure: soft-tissue surgery

INTERVENTIONS:
Procedure: Four-in-one procedure — "four-in-one" surgical technique centered on "tibial tuberosity osteotomy and proximal displacement"
  Arms: Study group
Procedure: soft-tissue surgery — traditional soft-tissue surgery
  Arms: Control group

SUMMARY:
Adult habitual dislocation of the patella is a common dislocation of the patella. The range of lesions is wide and the severity is high. Clinical diagnosis and treatment are difficult. In clinical work, misdiagnosis and treatment are not targeted at pathological mechanisms. This leads to irregular diagnosis and treatment, high failure rate and revision rate, and patients undergoing multiple operations. The project team developed a "four-in-one" surgical technique centered on "tibial tuberosity osteotomy and proximal displacement" in the preliminary research, which overcomes the disadvantages of traditional knee extension surgery and is suitable for adults. Early research Shows safe and effective clinical efficacy. The purpose of this application project is to take independent innovation of core surgical technology as the lead, adopt a two-way cohort study method, compare the clinical efficacy of the new "four-in-one" technology and traditional soft tissue surgery in the treatment of adult habitual patellar dislocation, and analyze and formulate adult habituation Comprehensive and systematic solutions for patella dislocation, relying on this scientific research project to conduct multi-center and large-sample clinical case studies, and evaluate the effectiveness and safety of independent innovative technologies through standardized medical research methods to improve the surgical treatment of adult habitual patella dislocation Success rate, reduce recurrence rate and failure rate, improve the level of clinical treatment of the disease, and finally put forward a special clinical diagnosis and treatment system for the disease in the international academic community.

ELIGIBILITY:
Inclusion Criteria:

* Patients with habitual dislocation of the patella over 14 years old
* agree to participate in the study

Exclusion Criteria:

* Combined with other knee ligament injuries
* recurrent patellar dislocation
* Skin and soft tissue conditions do not allow surgery

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Kujala score | 1 year postoperatively
  A functional score used to assess the knee function
quadriceps strength | 1 year postoperatively
  quantify the quadriceps strength using Biodex®

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhang, Study Director — Sports Medicine Service, Beijing Jishuitan hospital

IPD SHARING:
Plan to Share IPD: No